CLINICAL TRIAL: NCT04349059
Title: The Impact of a Plant-Based Diet Versus an Animal-Based Diet on Erectile Function in Healthy Men With Normal Erectile Function: The ERECTION Study
Brief Title: The Impact of Dietary Pattern on Erectile Function
Acronym: ERECTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Purjes Foundation (Unknown); The Greenbaum Foundation (Unknown); Nitric Oxide Innovations LLC (Industry); National Institutes of Health (NIH) (NIH); Dr. Irwin Goldstein (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-10465
Record Dates: First submitted 2020-03-27; First posted 2020-04-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction
Keywords: Diet; Erectile function; Plant-based; Animal-based
MeSH Terms: conditions — Erectile Dysfunction | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to randomization group and order of testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based arm (Active Comparator): The plant-based arm consists of 3 visits to the clinical research center, following a plant-based diet and using the Rigiscan™ device to measure the frequency, rigidity, and duration of nocturnal erections.
  Interventions: Other: Plant based diet
- Animal-based arm (Active Comparator): The animal-based arm consists of 3 visits to the clinical research center, following an animal- based diet and using the Rigiscan™ device to measure the frequency, rigidity, and duration of nocturnal erections.
  Interventions: Other: Animal based diet

INTERVENTIONS:
Other: Animal based diet — Food will be provided by Montefiore-Einstein Food Services
  Arms: Animal-based arm
Other: Plant based diet — Food will be provided by Montefiore-Einstein Food Services
  Arms: Plant-based arm

SUMMARY:
The goal of this study is to determine whether erectile function is impacted by dietary patterns in healthy men with normal erectile function.

DETAILED DESCRIPTION:
Visit 1:

After reviewing and signing consent, subjects will be screened for the study. Screening will consist of the following:

* Complete International Index of Erectile Function (IIEF) questionnaire.
* Record medical history, concomitant medications
* Measure height and weight, calculate BMI
* Vitals
* Draw blood for total testosterone, sex hormone binding globulin and Thyroid Stimulating Hormone
* Query subject regarding the presence of genital rash or lesions. Subjects will be asked, "do you have a rash or lesion on your penis or surrounding area?"

If the IIEF score is abnormal, subjects will be advised to contact their primary care provider.

Each subject will be contacted by phone with their blood results. If abnormal subject will be given the recommendation to contact his primary care provider.

If an abnormal finding is identified during screening, such as an abnormal STOP-bang score, subject will be given the recommendation to contact his primary care provider.

If the subject has no primary care provider, contact information for primary care will be given.

Subjects meeting inclusion and exclusion criteria will be randomized into the study, into either Sequence One or Sequence Two. Once enrolled, subjects will be asked to not modify their dietary habits throughout the duration of the study other than during the two evenings and two full days when food is provided (see below).

Sequence One:

Visit 2:

Subjects will return to the study center in the morning after having fasted (other than consuming water) since 11pm the night before. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be made. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

Subjects will be taught how to use the Rigiscan™ device. Subjects will receive one plant-based dinner (food will be provided by Montefiore-Einstein Food Services.) Subjects will then leave the study center and they will consume their usual diet until 5pm. For the rest of the evening until 11pm they will consume only the dinner provided. Water will be the only beverage allowed after 5pm. Dinner should be consumed at 8:30pm EST. Subjects will text pictures of everything they consume (eat or drink) after 5pm to Dr. Ostfeld or to a study representative and s/he will have text or verbal contact with the subject at least once that evening. That night, subjects will do a Rigiscan™ assessment overnight at their home. The time the subject goes to bed and the time the subject wakes up for the day should be recorded. The subject agrees to be in bed with Rigiscan™ on (other than for emergency or needed trips to the bathroom) for at least seven hours.

Visit 3 Subjects will return to the study center the morning after the Rigiscan™ assessment and bring the Rigiscan™ device with them. They will have been fasting other than drinking water since 11pm the night before. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be taken. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

Subjects will then receive one full day of plant-based meals (food will be provided by Montefiore-Einstein Food Services.) Subjects will be encouraged to eat breakfast at the study center after the initial anthropomorphic measures are made, saliva is obtained, and blood is drawn. Subjects will text pictures of all they consume during that day to Dr. Ostfeld and/or to a study representative and s/he will have text or verbal contact with the subject at least twice during that day. Dinner should be consumed at 8:30pm, EST. Subjects will fast other than water after 11pm. That night, subjects will do a Rigiscan™ assessment overnight at their home. Black coffee and/or tea is permitted only before noon. The time the subject goes to bed and the time the subject wakes up for the day should be recorded. The subject agrees to be in bed with Rigiscan™ on (other than for emergency or needed trips to the bathroom) for at least seven hours.

Visit 4 Subjects will return to the study center the morning after the Rigiscan™ assessment and bring the Rigiscan™ device with them. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be taken. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

There will then be a washout period for 8-12 days and subjects will be instructed to return to their usual dietary habits during this washout period. Number of days of the washout period will be recorded.

Visit 5 After the washout period, subjects will return to the study center in the morning after having fasted (other than consuming water) since 11pm the night before. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be taken. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

Subjects will receive one animal-based dinner (food will be provided by Montefiore-Einstein Food Services.) Subjects will then leave the study center and they will consume their usual diet until 5pm. For the rest of the evening until 11pm they will consume only the dinner provided. Water will be the only beverage consumed after 5pm. Dinner should be consumed at 8:30pm, EST. Subjects will text pictures of all they consume (eat or drink) after 5pm to Dr. Ostfeld or to a study representative and s/he will have text or verbal contact with the subject at least once that evening. Subjects will fast other than water after 11pm. That night, subjects will do a Rigiscan™ assessment overnight at their home. The time the subject goes to bed and the time the subject wakes up for the day should be recorded. The subject agrees to be in bed with Rigiscan™ on (other than for emergency or needed trips to the bathroom) for at least seven hours.

Visit 6 Subjects will return to the study center the morning after the Rigiscan™ assessment and bring the Rigiscan™ device with them. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be taken. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

Subjects will then receive one full day of animal-based meals (food will be provided by Montefiore-Einstein Food Services.) Subjects will be encouraged to eat breakfast at the study center after the initial anthropomorphic measures are made, saliva is obtained, and blood is drawn. Subjects will text pictures of all they consume during that day to Dr. Ostfeld and/or to a study representative and s/he will have text or verbal contact with the subject at least twice during that day. Dinner should be consumed at 8:30pm, EST. Subjects will fast other than water after 11pm. That night, subjects will do a Rigiscan™ assessment overnight at their home. Black coffee and/or tea is permitted only before noon. The time the subject goes to bed and the time the subject wakes up for the day should be recorded. The subject agrees to be in bed with Rigiscan™ on (other than for emergency or needed trips to the bathroom) for at least seven hours.

Visit 7 (End of Study) Subjects will return to the study center the morning after the Rigiscan™ assessment and bring the Rigiscan™ device with them. They will have been asked to not brush their teeth or use mouthwash and/or other breath fresheners that morning. Anthropomorphic and blood pressure and heart rate recordings will be taken. Saliva will be stored for NO measurement. Blood will be drawn and stored. Urine will be collected and stored.

Sequence Two:

Sequence Two is identical to Sequence One, except that the order of the plant-based and animal-based meals is reversed.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent and HIPAA authorization in English before any study procedures are conducted.
* Subject is taking no medical therapy other than: prn MDIs, medication(s) for anxiety, depression, and/or ADHD (these medications include, but are not limited to, SSRIs, SNRIs, Stimulants), no change in supplements if applicable.

The anxiety, depression, and/or ADHD will have been controlled (per report of subject) for the last 6 months.

* IIEF score greater or equal to 22
* Subject will have had penile-sexual intercourse (either vaginal or anal penetration) within 12 weeks of enrollment.
* Male aged 18-35 years old
* Lives within commuting distance of Montefiore Health System
* Subject's significant other (if applicable) agrees to support the subject during the study
* Subject agrees to photograph and share all items consumed/drunk during the dietary intervention
* Subject agrees to avoid all illicit drugs, NSAIDS, and alcohol for at least two days prior to Rigiscan™ recording and on the days and nights of Rigiscan™ recording
* Subject agrees to refrain from sexual activity for at least 24 hours prior to Rigiscan™ placement and to have no sexual activity on the days and nights of Rigiscan™ recording.
* Subject agrees to not view, read, or otherwise consume erotic or pornographic material for 24 hours prior to both the days and nights of Rigiscan™ recording and on the days and nights of Rigiscan™ recording.
* Subject agrees to not have an orgasm for 24 hours prior to both the days and nights of RigiscanTM recording and on the days and nights of Rigiscan™ recording.
* Subject agrees to come to Montefiore to undergo Rigiscan™ training
* Subject agrees to only consume/drink permitted food/beverages.
* Subject agrees to attend all in person visits at Montefiore, to begin fasting at 11pm the night before each visit, and to undergo all blood draws/salivary/other testing.
* Subject agrees to not use mouthwash or mouth rinses or intentionally spit for the entire duration of the study. Subjects will be asked to refrain from using mouthwash for at least 2 days prior to enrollment. Subject agrees to not brush his teeth in the morning of the day of each study visit. Tooth brushing is otherwise permissible.
* BMI <30, BMI >=18.5, weight >110 lbs.
* Subject agrees to comply with the study procedures and visits.
* Subject exercises for at least 15 minutes at least two times per week
* If exercise is done, subjects will exercise for the same amount of time and at a similar intensity each day of Rigiscan™ testing. Otherwise, no exercise will be performed on Rigiscan™ days.
* If enrolled, subjects agree to not modify their dietary habits throughout the duration of the study other than during the two evenings and two full days when food is provided.

Exclusion Criteria:

* Relevant dietary allergy
* Vegetarian or Vegan dietary pattern
* History of an eating disorder and/or food addiction
* Hypertension and or history of hypertension with or without medical treatment. Systolic blood pressure > 150mmHg and/or diastolic blood pressure >100mmHg on Visit one. Heart rate >99 on Visit one. Systolic blood pressure < 85mmHg and/or diastolic blood pressure < 50mmHg on Visit one. Heart rate < 35 on Visit one.
* BMI >=30, BMI <18.5, or weight <= 110lbs
* Known chronic medical disease other than non-inflammatory musculoskeletal disease, asthma, anxiety, depression, and/or ADHD.

Subjects who have had changes in the dosage or type of their medication(s) for anxiety, depression, and/or ADHD within 3 months of enrollment.

Subjects who have scheduled or planned medication and/or medication dose changes during the study period. These medication changes include the initiation of a new medication, discontinuation of a medication, modification of medication dose, and/or the route of administration of a medication.

Subjects who are taking benzodiazepines and/or beta blockers

* History of kidney disease or hyperkalemia
* Subject has received an investigational drug within 30 days prior to signing consent
* Erectile dysfunction
* Has any condition (e.g., psychiatric illness) or situation that, in the investigator's opinion, may confound the study results, or may interfere significantly with the patient's ability to adhere with study procedures
* Currently undergoing treatment for Peyronie's Disease
* Abnormal Testosterone or Thyroid Stimulating Hormone level
* Treated hypogonadism or hypothyroidism
* Planned travel during the study
* The subject is trans-gender
* History of substance abuse in the last 12 months
* Illicit drug use, smoking, or vaping within 4 weeks
* Upper respiratory illness within two weeks on screening
* If profession requires being on call, no overnight or on call duties during the study
* Subject reports any communicable skin or venereal disease
* Subject reports rash or lesion on the penis or surrounding area.
* STOP-Bang score > 2
* Having the diagnosis of Restless Leg Syndrome.
* Having insomnia as defined by: Subject with insomnia would have difficulty initiating or maintaining sleep (30 minutes or more at sleep initiation or 30 minutes or more to fall back asleep if wakes during the night). The above occurs at least 3 times per week for at least 1 month. Furthermore, there must be adequate opportunity for sleep and there must be associated morbidity (feels tired during the day). Definition based on: The International Classification of Sleep Disorders - Third Edition (ICSD-3), 2014.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent of time ≥70% erect during overnight sleep after 4 meals. | During overnight sleep directly after consuming the 4 meals.
  Total time (in minutes) when penile rigidity is ≥ 70% at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™).

SECONDARY OUTCOMES:
Percent of time ≥70% erect during overnight sleep after 1 meal. | During overnight sleep directly after consuming the 1 meal.
  Total time (in minutes) when penile rigidity is ≥70% at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™).
Erection events per hour during overnight sleep after 4 meals. | During overnight sleep directly after consuming the 4 meals.
  Total number of erection events lasting ≥5 minutes and with ≥70% rigidity at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™). This result will be reported as Events/hour.
Tumescence events per hour during overnight sleep after 4 meals. | During overnight sleep directly after consuming the 4 meals.
  Total number of tumescence events lasting ≥5 minutes and when penile circumference increases by ≥2cm at both the tip and the base of the penis compared to their respective baselines as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™). This result will be reported as Tumescence events/hour

OTHER OUTCOMES:
Heart rate | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing heart rate by dietary pattern at both time points (after overnight sleep after consuming the 1 meal and after overnight sleep after consuming the 4 meals) and compared to its respective baseline in beats/minute. Definition: In regard to the following anthropometric, vital sign, and laboratory data (blood, urine, and saliva) pre-specified outcomes included in this pre-specified outcomes section, at "both time points" is defined as in the sentence above and "respective baseline" refers to either visit 2 or visit 5, as visit 2 is the baseline for one dietary arm (plant or animal) and visit 5 is the baseline for the other dietary arm (plant or animal).
Blood Pressure | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing blood pressure by dietary pattern at both time points and compared to its respective baseline in mmHg
Weight | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing weight by dietary pattern at both time points and compared to its respective baseline
Fibrinogen | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
D-dimer | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in ng/mL
Total cholesterol | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
HDL cholesterol | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
HDL efflux capacity | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline.
LDL cholesterol | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Triglyceride | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Oxidized LDL cholesterol | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in U/L
Free Fatty Acids | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in micromoles
Myeloperoxidase | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in ug/L
Factor VII | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in percentage.
lysolecithin | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/mL
Apolipoprotein B | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Omega 3 index | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in percentage of erythrocyte fatty acid
Lipoprotein-associated phospholipase-A2 (Lp PLA2) activity | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in nmol/min/mL
Lipoprotein (a) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in nmol/L
Homocysteine | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
methylmalonic acid (MMA) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
Asymmetric Dimethylarginine (ADMA) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
symmetric dimethylarginine (SDMA) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Total testosterone | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Sex Hormone Binding Globulin | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in nmol/L
cystatin C | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
remnant cholesterol particles | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
uric acid | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
interleukin 1 | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in pg/mL
interleukin 6 | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in pg/mL
hsCRP | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/L
Blood Urea Nitrogen (BUN) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
Carbon Dioxide (CO2) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mmol/L
creatinine | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
glucose | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
serum chloride | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in meq/L
serum potassium | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in meq/L
serum sodium | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in meq/L
alanine aminotransferase (ALT) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in units/L
aspartate aminotransferase (AST) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in units/L
estimated glomerular filtration rate (eGFR) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mL/min/1.73m2
vitamin c | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/dL
reduced glutathione | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
superoxide dismutase | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in ng/mL
vitamin e | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/L
selenium | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in ng/mL
malondialdehyde | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
non coding RNA | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in copies/mL
micro RNA | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in copies/mL
Lnc RNA | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in copies/mL
trimethylamine-N-oxide (TMAO) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in umol/L
phenylacetylglutamine (PAG) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in uM (micrometers)
Comparing urine albumin-to-creatinine ratio (UACR) | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in mg/g
Comparing salivary nitrite level as a correlate of plasma nitric oxide (NO) level | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in micromoles/L
Comparing salivary nitrate level in as a correlate of plasma nitric oxide (NO) level | Time zero (Visit 2, ~1-21 days after screen), at ~24 hours after time zero (Visit 3), at ~48 hours after time zero (Visit 4), after 8-12 day washout (Visit 5), at ~24 hours after 8-12 day washout (Visit 6), at ~48 hours after 8-12 day washout (Visit 7)
  Comparing it at both time points by dietary pattern and compared to its respective baseline in micromoles/L
Percent of time ≥50% erect during overnight sleep after 4 meals. | During overnight sleep directly after consuming the 4 meals.
  Total time (in minutes) when penile rigidity is ≥50% at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™).
Percent of time ≥50% erect during overnight sleep after 1 meal. | During overnight sleep directly after consuming the 1 meal.
  Total time (in minutes) when penile rigidity is ≥50% at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™).
Erection events per hour during overnight sleep after 1 meal. | During overnight sleep directly after consuming the 1 meal.
  Total number of erection events lasting ≥5 minutes and with ≥70% rigidity at both the tip and the base of the penis as measured by Rigiscan™ during overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™). This result will be reported as Events/hour.
Tumescence events per hour during overnight sleep after 1 meal. | During overnight sleep directly after consuming the 1 meal.
  Total number of tumescence events lasting ≥5 minutes and when penile circumference increases by ≥2cm at both the tip and the base of the penis compared to their respective baselines as measured by Rigiscan™ during overnight sleep, divided by the total time (in minutes) of overnight sleep. Overnight sleep is defined as the time in minutes from the onset of the first nocturnal erection to the end of the last nocturnal erection (as measured by Rigiscan™). This result will be reported as Tumescence events/hour.
Percent of time ≥70% erect during overnight sleep after 4 meals versus after 1 meal by dietary pattern. | During overnight sleep directly after consuming the 4 meals versus overnight sleep directly after consuming the 1 meal by dietary pattern, for each dietary pattern.
  This outcome will evaluate whether a difference is present in the percent of time ≥70% erect during overnight sleep (as defined in outcomes above) directly after consuming the 4 meals versus directly after consuming the 1 meal by dietary pattern, for each dietary pattern. (e.g. is there a greater percentage of time ≥70% erect on the second night versus the first night when consuming the plant-based diet?).
Percent of time ≥50% erect during overnight sleep after 4 meals versus after 1 meal by dietary pattern. | During overnight sleep directly after consuming the 4 meals versus overnight sleep directly after consuming the 1 meal by dietary pattern, for each dietary pattern.
  This outcome will evaluate whether a difference is present in the percent of time ≥50% erect during overnight sleep (as defined in outcomes above) directly after consuming the 4 meals versus directly after consuming the 1 meal by dietary pattern, for each dietary pattern. (e.g. is there a greater percentage of time ≥50% erect on the second night versus the first night when consuming the plant-based diet?).
Tumescence events per hour during overnight sleep after 4 meals versus after 1 meal by dietary pattern. | During overnight sleep directly after consuming the 4 meals versus overnight sleep directly after consuming the 1 meal by dietary pattern, for each dietary pattern.
  This outcome will evaluate whether a difference is present in the total number of tumescence events per hour (as defined in outcomes above) directly after consuming the 4 meals versus directly after consuming the 1 meal by dietary pattern, for each dietary pattern. (e.g. is there a greater of tumescence events per hour on the second night versus the first night when consuming the plant-based diet?).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ostfeld, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, Department of Medicine, Division of Cardiology, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Nehra A. Erectile dysfunction and cardiovascular disease: efficacy and safety of phosphodiesterase type 5 inhibitors in men with both conditions. Mayo Clin Proc. 2009 Feb;84(2):139-48. doi: 10.4065/84.2.139. PMID 19181648
- [Background] Thompson IM, Tangen CM, Goodman PJ, Probstfield JL, Moinpour CM, Coltman CA. Erectile dysfunction and subsequent cardiovascular disease. JAMA. 2005 Dec 21;294(23):2996-3002. doi: 10.1001/jama.294.23.2996. PMID 16414947
- [Background] Vogel RA, Corretti MC, Plotnick GD. Effect of a single high-fat meal on endothelial function in healthy subjects. Am J Cardiol. 1997 Feb 1;79(3):350-4. doi: 10.1016/s0002-9149(96)00760-6. PMID 9036757
- [Background] Ong PJ, Dean TS, Hayward CS, Della Monica PL, Sanders TA, Collins P. Effect of fat and carbohydrate consumption on endothelial function. Lancet. 1999 Dec 18-25;354(9196):2134. doi: 10.1016/s0140-6736(99)03374-7. PMID 10609824
- [Background] Esposito K, Nappo F, Giugliano F, Giugliano G, Marfella R, Giugliano D. Effect of dietary antioxidants on postprandial endothelial dysfunction induced by a high-fat meal in healthy subjects. Am J Clin Nutr. 2003 Jan;77(1):139-43. doi: 10.1093/ajcn/77.1.139. PMID 12499333
- [Background] Shimabukuro M, Chinen I, Higa N, Takasu N, Yamakawa K, Ueda S. Effects of dietary composition on postprandial endothelial function and adiponectin concentrations in healthy humans: a crossover controlled study. Am J Clin Nutr. 2007 Oct;86(4):923-8. doi: 10.1093/ajcn/86.4.923. PMID 17921366
- [Background] Sakakibara S, Murakami R, Takahashi M, Fushimi T, Murohara T, Kishi M, Kajimoto Y, Kitakaze M, Kaga T. Vinegar intake enhances flow-mediated vasodilatation via upregulation of endothelial nitric oxide synthase activity. Biosci Biotechnol Biochem. 2010;74(5):1055-61. doi: 10.1271/bbb.90953. Epub 2010 May 7. PMID 20460711
- [Background] Esposito K, Ciotola M, Giugliano F, De Sio M, Giugliano G, D'armiento M, Giugliano D. Mediterranean diet improves erectile function in subjects with the metabolic syndrome. Int J Impot Res. 2006 Jul-Aug;18(4):405-10. doi: 10.1038/sj.ijir.3901447. Epub 2006 Jan 5. PMID 16395320
- [Background] Wing RR, Rosen RC, Fava JL, Bahnson J, Brancati F, Gendrano Iii IN, Kitabchi A, Schneider SH, Wadden TA. Effects of weight loss intervention on erectile function in older men with type 2 diabetes in the Look AHEAD trial. J Sex Med. 2010 Jan;7(1 Pt 1):156-65. doi: 10.1111/j.1743-6109.2009.01458.x. Epub 2009 Aug 17. PMID 19694925
- [Background] Gupta BP, Murad MH, Clifton MM, Prokop L, Nehra A, Kopecky SL. The effect of lifestyle modification and cardiovascular risk factor reduction on erectile dysfunction: a systematic review and meta-analysis. Arch Intern Med. 2011 Nov 14;171(20):1797-803. doi: 10.1001/archinternmed.2011.440. Epub 2011 Sep 12. PMID 21911624
- [Background] Cassidy A, Franz M, Rimm EB. Dietary flavonoid intake and incidence of erectile dysfunction. Am J Clin Nutr. 2016 Feb;103(2):534-41. doi: 10.3945/ajcn.115.122010. Epub 2016 Jan 13. PMID 26762373
- [Background] Yaman O, Tokath Z, Inal T, Anafarta K. Effect of sildenafil on nocturnal erections of potent men. Int J Impot Res. 2003 Apr;15(2):117-21. doi: 10.1038/sj.ijir.3900978. PMID 12789391
- [Background] Corbin JD, Francis SH. Cyclic GMP phosphodiesterase-5: target of sildenafil. J Biol Chem. 1999 May 14;274(20):13729-32. doi: 10.1074/jbc.274.20.13729. No abstract available. PMID 10318772
- [Background] Greenstein A, Chen J, Salonia A, Sofer M, Matzkin H, Montorsi F. Does sildenafil enhance quality of nocturnal erections in healthy young men? A NPT-RigiScan study. J Sex Med. 2004 Nov;1(3):314-7. doi: 10.1111/j.1743-6109.04045.x. PMID 16422962
- [Background] Burris AS, Banks SM, Sherins RJ. Quantitative assessment of nocturnal penile tumescence and rigidity in normal men using a home monitor. J Androl. 1989 Nov-Dec;10(6):492-7. doi: 10.1002/j.1939-4640.1989.tb00148.x. PMID 2621154
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880